CLINICAL TRIAL: NCT05175781
Title: Dexmedetomidine Versus Ketamine to Facilitate Non-invasive Ventilation After Blunt Chest Trauma
Brief Title: Sedation for Non-invasive Ventilation in Blunt Chest Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Huda Fahmy Mahmoud, PhD, Director, anaesthesia and ocu department, Principal Investigator, Clinical Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 494/12/20
Record Dates: First submitted 2021-11-07; First posted 2022-01-04 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Chest Trauma
Keywords: Sedation - noninvasive ventilation-ketamine- dexmedetomidine
MeSH Terms: conditions — Thoracic Injuries | interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dexmedetomidine (Active Comparator): patients will receive two NIV sessions during which intravenous continuous infusion of dexmedetomidine will be given.
  The infusion was initiated 60 min prior to NIV at the same rate for all treatments, corresponding to 0.7 mcg/kg/h of dexmedetomidine without a loading dose. Dexmedetomidine will then titrate by 0.2 mcg/kg/h every 60 min (up to a maximum dose of 1.3 mcg/kg/h) to maintain a RASS score between 0 and 3. A 6-h washout period was observed between two NIV sessions accounting for 1-h contextual half-life of dexmedetomidine. Patients received neither tested drug nor NIV during this 6-h interval.
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Ketamine (Active Comparator): patients will receive two NIV sessions during which intravenous continuous infusion of ketamine will be given.
  The infusion was initiated 60 min prior to NIV at the same rate for all treatments, infusion of ketamine will be at the dose of 0.20 mg/kg/h (or 3.3 mg/kg/min). to maintain a RASS score between 0 and 3. A 6-h washout period was observed between two NIV sessions . Patients received neither tested drug nor NIV during this 6-h interval.
  Following the start of the infusion, the patient could have a morphine dose if the 10-cm Visual Analog Scale (VAS) exceeded 3.
  Interventions: Drug: Ketamine Hydrochloride
- Placebo (Placebo Comparator): patients will receive two NIV sessions during which intravenous continuous infusion of placebo (0.9% sodium chloride solution) will be given.
  The infusion was initiated 60 min prior to NIV at the same rate for all treatments, corresponding to 0.7 mcg/kg/h of dexmedetomidine without a loading dose. will then titrate by 0.2 mcg/kg/h every 60 min (up to a maximum dose of 1.3 mcg/kg/h) to maintain a RASS score between 0 and 3. A 6-h washout period was observed between two . Patients received neither tested drug nor NIV during this 6-h interval.
  Following the start of any infusion, the patient could have a morphine dose if the 10-cm Visual Analog Scale (VAS) exceeded 3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — is a sympatholytic drug that acts as an agonist of α2-adrenergic receptors in certain parts of the brain.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Ketamine Hydrochloride — Ketamine is an NMDA receptor antagoni
  Other Names: Ketalar
  Arms: Ketamine
Drug: Placebo — Normal saline
  Other Names: Nacl .9%
  Arms: Placebo

SUMMARY:
Effectiveness of sedation using dexmedetomidine and ketamine to facilitate non-invasive ventilation sessions which improve overall outcome after blunt chest trauma

DETAILED DESCRIPTION:
Chest trauma remains an issue for health services for both severe and apparently mild trauma management. Severe chest trauma is associated with high mortality and is considered liable for 25% of mortality in multiple traumas. Moreover, mild trauma is also associated with significant morbidity especially in patients with preexisting conditions. Thus, whatever the severity, a fast-acting strategy must be organized.

Blunt traumas are commonly secondary to motor vehicle accidents, falls, and crush or blast injuries. They are the most common type of thoracic trauma, accounting for over 90%, and are often associated with rib fractures, haemothorax, pneumothorax, and pulmonary contusions.

In order to improve the prognosis of patients with severe chest trauma, early and continuous application of non-invasive mechanical ventilation (NIV) can indeed reduce the need for intubation and shorten intensive care unit length-of-stay Among different mechanisms, the early use of positive end-expiratory pressure after chest trauma, when feasible, seems mandatory to optimize oxygenation and improve clinical outcomes. Indeed, interventions aimed at preventing acute respiratory distress syndrome (ARDS) after chest trauma carry the greatest potential to reduce the substantial morbidity, mortality, and resource utilization associated with this syndrome.

Notably, pain control seems a crucial endpoint in our success to deliver non-invasive ventilation to patients with chest trauma, when feasible as a pivotal component of patient care after chest trauma, along with non-invasive ventilation. In this context, the role of intensivist doctors is thus to provide optimal control of chest wall pain, respiratory comfort, agitation, and anxiety as a prerequisite to reduce the incidence of NIV failure in this trauma population.

In this context, dexmedetomidine could be an alternative to improve NIV tolerance. Dexmedetomidine is a short-acting alpha-2 adrenoreceptor agonist that provides sedation and analgesia with no significant respiratory depression and a reduced risk of delirium.

Ketamine has several advantages compared with conventional sedatives such as preserving pharyngeal and laryngeal protective reflexes, lowering airway resistance, increasing lung compliance, and being less likely to produce respiratory depression. It causes sympathetic stimulation, which is also unlike other sedatives and analgesics.

However, no studies have estimated the superiority of dexmedetomidine or Ketamine to improve analgesia and non-invasive ventilation tolerance in patients with blunt chest

The patients will be randomly allocated into 3 groups, the allocation of the treatment order will determine by means of a computer-generated random table.

Group C: will receive placebo infusion (0.9% sodium chloride solution) Group D: will receive dexmedetomidine infusion Group K: will receive ketamine infusion

ELIGIBILITY:
Inclusion Criteria:

All blunt chest trauma patients with:

* More than 3 rib fractures, pulmonary contusion,
* hypoxemia or hypercapnia, or respiratory rate 20/ min despite an optimized intravenous analgesia ( paracetamol 1gm i.v. 6hourly and ketolac 30mg i.v. 8 hourly)
* No indication of mechanical ventilation

Exclusion Criteria:

* Patients < 18 years old,
* admitted under mechanical ventilation
* admitted more than 24 h after trauma or from another hospital,
* patients with less than 3 ribs fractures
* patients did not receive CT-scan
* Patients in whom alpha-2 agonists or ketamine are contraindicated
* Patients who will require an intubation during the study period for a life-threatening condition or emergency surgery or agitation as defined by a Richmond Agitation Sedation Scale (RASS) score higher than +2 will also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Duration of non-invasive ventilation (NIV) session | 8 hours
  duration that patient can withhold NIV comfortably

SECONDARY OUTCOMES:
Richmond agitation sedation score (RASS) | 8 hours
  The hourly measurements by nurses of RASS score for pain and respiratory discomfort during each NIV session.
Visual analogue scale | 8 hours
  the hourly measurements of self-rated 10-cm VAS for pain during each NIV session.
length of ICU stay | 8 days
  Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- AHU, Aswān, Egypt

REFERENCES:
- [Background] Deletombe B, Trouve-Buisson T, Godon A, Falcon D, Giorgis-Allemand L, Bouzat P, Bosson JL, Payen JF. Dexmedetomidine to facilitate non-invasive ventilation after blunt chest trauma: A randomised, double-blind, crossover, placebo-controlled pilot study. Anaesth Crit Care Pain Med. 2019 Oct;38(5):477-483. doi: 10.1016/j.accpm.2019.06.012. Epub 2019 Jul 15. PMID 31319192
- [Background] Bouzat P, Raux M, David JS, Tazarourte K, Galinski M, Desmettre T, Garrigue D, Ducros L, Michelet P; Expert's group; Freysz M, Savary D, Rayeh-Pelardy F, Laplace C, Duponq R, Monnin Bares V, D'Journo XB, Boddaert G, Boutonnet M, Pierre S, Leone M, Honnart D, Biais M, Vardon F. Chest trauma: First 48hours management. Anaesth Crit Care Pain Med. 2017 Apr;36(2):135-145. doi: 10.1016/j.accpm.2017.01.003. Epub 2017 Jan 16. PMID 28096063
- [Background] Erstad BL, Patanwala AE. Ketamine for analgosedation in critically ill patients. J Crit Care. 2016 Oct;35:145-9. doi: 10.1016/j.jcrc.2016.05.016. Epub 2016 May 25. PMID 27481750
- [Background] Weerink MAS, Struys MMRF, Hannivoort LN, Barends CRM, Absalom AR, Colin P. Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine. Clin Pharmacokinet. 2017 Aug;56(8):893-913. doi: 10.1007/s40262-017-0507-7. PMID 28105598
- [Background] Jabaudon M, Blondonnet R, Constantin JM. ARDS in patients with chest trauma: Better safe than sorry. Anaesth Crit Care Pain Med. 2019 Jun;38(3):221-222. doi: 10.1016/j.accpm.2019.04.006. No abstract available. PMID 31076142
- [Background] Mion G, Villevieille T. Ketamine pharmacology: an update (pharmacodynamics and molecular aspects, recent findings). CNS Neurosci Ther. 2013 Jun;19(6):370-80. doi: 10.1111/cns.12099. Epub 2013 Apr 10. PMID 23575437
- [Background] Hoy SM, Keating GM. Dexmedetomidine: a review of its use for sedation in mechanically ventilated patients in an intensive care setting and for procedural sedation. Drugs. 2011 Jul 30;71(11):1481-501. doi: 10.2165/11207190-000000000-00000. PMID 21812509